CLINICAL TRIAL: NCT02306902
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioequivalence Study Comparing Fenofibrate Capsule 130 mg of Ohm Laboratories Inc., USA (A Subsidiary of Ranbaxy Pharmaceuticals Inc., USA) With Antara® Capsule 130 mg (Containing Fenofibrate 130 mg) of Oscient Pharmaceutical Corporation, USA in Healthy, Adult, Male Human Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Fenofibrate Capsules, 130 mg Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 243_FENOF_09
Record Dates: First submitted 2014-11-24; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Fenofibrate Capsules, USP 130 mg
  Interventions: Drug: fenofibrate
- Reference (Active Comparator): ANTARA® (fenofibrate) Capsules 130 mg
  Interventions: Drug: ANTARA® (fenofibrate)

INTERVENTIONS:
Drug: fenofibrate — 130mg, Capsules
  Arms: Test
Drug: ANTARA® (fenofibrate) — 130mg, Capsules
  Arms: Reference

SUMMARY:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioequivalence study comparing Fenofibrate capsules, USP 130 mg manufactured by Ohm Laboratories Inc, NJ 08901 with ANTARA® (fenofibrate) capsules 130 mg manufactured by Ethypharm Industries Saint Cloud, France for Oscient Pharmaceuticals Corp. Waltham, MA 02451 in healthy, adult, male, human subjects under fed condition.

DETAILED DESCRIPTION:
The subjects were subjected to breath test for alcohol and test for drugs of abuse (opioids and cannabinoids) in urine prior to admission in each period.

Following an overnight fast of at least 10 hour, a high-fat high calorie breakfast was served to the study subjects. Thirty minutes after start of this breakfast, a single oral dose of fenofibrate capsules 130 mg of either test or reference formulation was administered during each period of the study, along with 240 mL of drinking water at ambient temperature under low light condition and under supervision of trained study personnel.

Blood samples were collected at pre-dose and at 1.000, 2.000, 3.000, 4.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 7.500, 8.000, 8.500, 9.000, 9.500, 10.000, 11.000, 12.000, 16.000, 24.000, 36.000, 48.000, 72.000 and 96.000 hours post dose in each period under low light condition. The pre-dose blood samples in each period were collected in duplicate (2 x 5 mL), within a period of 1.5 hour before dosing. Post-dose samples were generally collected within 2 minutes of the scheduled time.

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis at screening). Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who met the following criteria were included in the study

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance
* Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
* Had a non-vegetarian dietary habit.

Exclusion Criteria:

* Subject had history of hypersensitivity to fenofibrate or any related drug or to any other drug.
* Subjects with history of hepatic or severe renal dysfunction, including primary biliary cirrhosis.
* Subjects with history of unexplained persistent liver function abnormality.
* Subjects with history of preexisting gallbladder disease.
* Subject had history of myalgia, muscle tenderness or weakness or myopathy
* Subject had any evidence of organ dysfunction or any clinically significant deviation from the normal in physical or clinical determinations.
* Clinically abnormal ECG or Chest X-ray, or hematological and biochemical parameters which was/were outside acceptable limits and was judged clinically significant by investigator.
* Investigations with blood samples of the subject showed presence of disease markers of HIV 1 or 2, Hepatitis B or C Viruses of syphilis infection.
* Investigations with urine samples of the subject showed clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4 /HPF), glucose (Positive) or Protein (Positive).
* Subject had history of serious medical illnesses including but not limited to gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes, glaucoma, any serious, potentially life-threatening illness.
* Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that might impair the ability to provide, written informed consent.
* Subject was a regular smoker, who smoked 10 or more cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* Subject had history of drug dependence or excessive alcohol intake on a habitual basis or has difficulty in abstaining for the duration of each study period.
* Use of any regular medication (OTC or prescription) or any drug metabolizing enzyme within 30 days prior to Day 1 of this study.
* Subject had participated in a clinical trial within 12 weeks preceding admission of this study (except for the subjects who dropout/withdrawn from the previous study prior to period I dosing).
* Subject had donated and/or lost more than 350 mL of blood in the past 3 months, including blood loss in this study.
* Consumption of alcohol for 48 hours prior to admission.
* Consumption of grapefruit juice and or grape fruit supplements containing products for 48 hours prior to admission.
* Subject had problem(s) in complying with the study protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of fenofibric acid | 0-96 hrs
Peak Plasma Concentration (Cmax) of fenofibric acid | 0-96 hrs

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm